CLINICAL TRIAL: NCT01126216
Title: Randomised Phase-III-trial of Simultaneous Radiochemotherapy (RCT) of Locally Advanced Head and Neck Cancer in the Stages III and IV A-B: Comparing Dose Reduced Radiotherapy (63,6 Gy) With Paclitaxel/Cisplatin to Standard Radiotherapy (70,2 Gy) With 5-Fluorouracil/Cisplatin
Brief Title: Reduced Radiotherapy With Pac/Cis vs Standard Radiotherapy With 5-FU/Cis in Locally Advanced Head and Neck Cancer
Acronym: Paccis-RCT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After an Interims analysis the Data Safety Monitoring board recommended this because no significant difference between the two arms was seen and was not expected with an reasonable recruitment of patients.
  No interruptions of the trial were made.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Paccis-RCT_2005; 2005-003484-23 (EudraCT Number); 107028 (Other Grant/Funding Number: Deutsche Krebshilfe e. V.)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer
Keywords: Radiochemotherapy; head and neck cancer; Paclitaxel; Cisplatin; 5-FU
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced RT + Pacitaxel/Cisplatin (Experimental): 63,6 Gy accelerated hyperfractionated radiotherapy with Paclitaxel (20mg/m^2/d) on days 2, 5, 8, 11 and 25, 30, 33, 36) and Cisplatin (20mg/m^2/d) on days 1-4 and 29-32, followed by a salvage operation or neck dissection if there is persisting tumor
  Interventions: Drug: Paclitaxel/Cisplatin; Radiation: Reduced RT
- Standard RT + 5-Fluorouracil/Cisplatin (Active Comparator): 70,6 Gy accelerated hyperfractionated radiotherapy with 5-Fluorouracil(600mg/m^2/d) on days 1-5 and 29-33) and Cisplatin (20mg/m^2/d) on days 1-5 and 29-33, followed by a salvage operation or neck dissection if there is persisting tumor
  Interventions: Drug: 5-FU/Cisplatin; Radiation: Standard RT

INTERVENTIONS:
Drug: Paclitaxel/Cisplatin — Experimental: Paclitaxel (20mg/m^2/d) on days 2, 5, 8, 11 and 25, 30, 33, 36) and Cisplatin (20mg/m^2/d) on days 1-4 and 29-32,
  Arms: Reduced RT + Pacitaxel/Cisplatin
Radiation: Reduced RT — Experimental: 63,6 Gy accelerated hyperfractionated radiotherapy
  Arms: Reduced RT + Pacitaxel/Cisplatin
Drug: 5-FU/Cisplatin — Active Comparator: 5-Fluorouracil(600mg/m^2/d) on days 1-5 and 29-33) and Cisplatin (20mg/m^2/d) on days 1-5 and 29-33
  Arms: Standard RT + 5-Fluorouracil/Cisplatin
Radiation: Standard RT — Active Comparator: 70,6 Gy accelerated hyperfractionated radiotherapy
  Arms: Standard RT + 5-Fluorouracil/Cisplatin

SUMMARY:
Reduced RT with Pac/Cis vs. standard RCT with 5-FU/Cis

DETAILED DESCRIPTION:
Standard treatment for patients with advanced, unresectable head and neck cancer is a platin-based simultaneous radiochemotherapy (RCT) (Pignon JP et al., Lancet 2000;355:949-955). However, irradiation dose is still debatable regarding local tumor control and late toxicity. Moreover, it is still unclear which combination of different drugs might be more effective.

In recent years, new drugs have been introduced in the field of head and neck cancer. The Taxanes, namely Docetaxel and Paclitaxel, have been investigated in several phase I/II-studies, and showed promising results concerning locoregional control rates and survival data. The RTOG 97-03 trial (Garden et al., J Clin Oncol 2004; 22:2856-64) compared a RCT either with Cisplatin/5-FU or Cisplatin/Paclitaxel. In this phase II-study an improvement of local tumor control and disease free survival of 15-20% in favour of the Cisplatin/Paclitaxel treatment arm was seen.

Therefore, our phase III-trial compares a standard RCT (70.6 Gy) with Cisplatin/5-FU to a RCT with Cisplatin/Paclitaxel and reduced irradiation dose (63.6 Gy). Primary endpoint is to proof superiority of the experimental Cisplatin/Paclitaxel treatment arm concerning disease-free-survival. Secondary endpoints are locoregional tumor control, overall survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, locally advanced stage III-IV A-B (UICC 2002) primary squamous cell carcinoma of the oral cavity, the oropharynx, the hypopharynx, the supraglottic larynx
* Age ≥ 18
* Written informed consent for the participation in the clinical trial

Exclusion Criteria:

* Inadequate hepatic function: Bilirubin > 2,0 mg/dl, SGOT, SGPT, AP, Gamma-GT > 3 x ULN
* Inadequate bone marrow function: leukocytes < 3,5 x 10^9/l, platelets < 100 x 10^9/l or neutrophils < 1,5 x 10^9/l
* Serum creatinine > 1,5 mg/dl, creatinine clearance < 60ml/min
* Uncontrolled severe somatic or psychological disease: e.g. unstable angina pectoris; myocardial infarction during the last 6 months; significant cardial rhythm disorders; apoplexy; high grade stenosis of the carotis; neurological or psychiatric disorders including convulsive disorders; dementia; psychosis; active uncontrolled infection or sepsis; liver cirrhosis; Child stage B,C; severe liver function disorders; marginal changes in the blood count; severe kidney damage; HIV-infection
* Acute infections
* Fertile women without adequate contraception during and up to 6 months after therapy (the method of contraception has to be high effective as described in the Note for guidance on non-clinical safety studies for the conduct of human clinical trials for pharmaceuticals (CPMP/ICH/286/95 mod) and it has to be discussed with the investigator)
* Pregnant or breast feeding women
* Men, who are not willing to use adequate contraception during and up to 6 months after therapy, that is discussed with the investigator
* ECOG-Status > 1
* Reduced hearing function (especially higher frequencies)
* Exsiccosis
* Neuropathy, caused by cisplatin
* Concurrent malignancies, with exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma or the cervix
* Prior radiotherapy of the neck or chemotherapy
* Distant metastasis
* Recurrent carcinoma in the head and neck region
* Prior neck-dissection or surgical intervention exceeding an exploratory excision
* Known intolerance to 5-Fluorouracil
* Known deficit of Dihydropyrimidine dehydrogenase (DPD)
* Simultaneous therapy with Brivudin or other inhibitors of DPD
* Known intolerance to Cisplatin or other substances that contain platin
* Known intolerance to Paclitaxel or one of the included substances, especially to Poly(oxyethylene)Rhizinusöl/Macrogolglycerol ricinoleate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
Distant metastasis free survival | 3 years
Local control | 3 years
Acute and Late Toxicity | 4 years
Life Quality | 4 years
HPV/p16-Status | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, MD, Study Director — Strahlenklinik, Universitätsklinikum Erlangen
Locations (13):
- Germany (13):
  - Klinikum Coburg, Strahlentherapie, DiaCura, Coburg
  - Universitätsklinikum Düsseldorf, Klinik und Poliklinik für Strahlentherapie und Radiologische Onkologie, Düsseldorf
  - Universitätsklinikum Erlangen, Strahlenklinik, Erlangen
  - Universitätsklinikum Frankfurt, Klinik für Strahlentherapie und Radioonkologie, Frankfurt/M.
  - Klinikum am Eichert, Praxis für Strahlentherapie und Klinik für Radioonkologie, Göppingen
  - Universitätsklinikum des Saarlandes, Klinik für Strahlentherapie und Radioonkologie,, Homburg/Saar
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Klinik und Poliklinik für Hals-Nasen- und Ohrenkranke, Lübeck
  - Kliniken Maria Hilf GmbH Mönchengladbach, Klinik für Strahlentherapie, Mönchengladbach
  - Klinikum München Pasing und Perlach, Klinik für HNO, München
  - Brüderkrankenhaus st. Josef Paderborn, Klinik für Strahlentherapie, Paderborn
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Strahlentherapie, Regensburg
  - Klinikum St. Elisabeth Straubing, Klinik für Hals-Nasen-Ohren-Heilkunde, Straubing
  - MVZ am Klinikum Mutterhaus der Borrmäerinnen, Strahlentherapie, Trier

REFERENCES:
- [Derived] Fietkau R, Hecht M, Hofner B, Lubgan D, Iro H, Gefeller O, Rodel C, Hautmann MG, Kolbl O, Salay A, Rube C, Melchior P, Breinl P, Krings W, Gripp S, Wollenberg B, Keerl R, Schreck U, Siekmeyer B, Grabenbauer GG, Balermpas P; PacCis-Study Group. Randomized phase-III-trial of concurrent chemoradiation for locally advanced head and neck cancer comparing dose reduced radiotherapy with paclitaxel/cisplatin to standard radiotherapy with fluorouracil/cisplatin: The PacCis-trial. Radiother Oncol. 2020 Mar;144:209-217. doi: 10.1016/j.radonc.2020.01.016. Epub 2020 Feb 7. PMID 32044419